CLINICAL TRIAL: NCT00482638
Title: Study of Safety, Tolerability and Efficacy of MK0493 in Obese Patients (0493-008)(COMPLETED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0493-008; 2007_571
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — N-1-(2-(1-(tert-butyl-4-(2,4-difluorophenyl)pyrrolidin-3-yl)-5-chlorophenyl)ethyl)acetamide

INTERVENTIONS:
Drug: MK0493

SUMMARY:
To assess the effect of MK0493 on body weight, blood pressure, mood, and appetite.

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 21 and 65 years
* Patient is able to read and understand and complete study questionnaires
* Patient is not pregnant or breast-feeding and does not plan to become pregnant for the duration of the study and post-study follow-up period

Exclusion Criteria:

* Patient has a history of significant psychiatric disorder (such as major depression, bipolar disorder, bulimia, or anorexia nervosa
* Patient is HIV positive as determined by medical history
* Patient has undergone surgical treatment for obesity
* Patient plans to consume more than two 8 ounce glasses of grapefruit juice per day during the study
* Patient participated in another clinical study involving an investigational drug) within 3 months prior to Visit 1
* Patient is currently a heavy consumer of alcohol (>2 drinks per day or >14 drinks per week [1 drink is defined as 2 oz hard alcohol, 5 oz wine, 12 oz beer], or uses (including recreational use) any illicit drugs, or has a history of drug or alcohol abuse

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-05-12 (Actual); Primary Completion 2004-10-29 (Actual); Study Completion 2004-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Krishna R, Gumbiner B, Stevens C, Musser B, Mallick M, Suryawanshi S, Maganti L, Zhu H, Han TH, Scherer L, Simpson B, Cosgrove D, Gottesdiener K, Amatruda J, Rolls BJ, Blundell J, Bray GA, Fujioka K, Heymsfield SB, Wagner JA, Herman GA. Potent and selective agonism of the melanocortin receptor 4 with MK-0493 does not induce weight loss in obese human subjects: energy intake predicts lack of weight loss efficacy. Clin Pharmacol Ther. 2009 Dec;86(6):659-66. doi: 10.1038/clpt.2009.167. Epub 2009 Sep 9. PMID 19741604